CLINICAL TRIAL: NCT01844297
Title: Efficacy and Safety of Tenofovir Disoproxil Fumarate Plus Lamivudine Plus Efavirenz Regimen as First-line Antiretroviral Therapy for ART-naive Chinese Patients With HIV-1 Infection
Brief Title: Efficacy and Safety of Tenofovir Plus Lamivudine Plus Efavirenz Regimen as First-line Antiretroviral Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, LI Taisheng, director of the Department of Infectious Disease, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACT1215
Record Dates: First submitted 2012-08-24; First posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: AIDS/HIV PROBLEM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TDF+3TC+EFV (Other)
  Interventions: Drug: TDF+3TC+EFV

INTERVENTIONS:
Drug: TDF+3TC+EFV

SUMMARY:
This study aims to evaluate the safety and effectiveness of the tenofovir disoproxil fumarate (TDF) + lamivudine (3TC) + efavirenz (EFV) regimen in antiretroviral therapy (ART)-naive Chinese HIV/AIDS patients.

DETAILED DESCRIPTION:
This study is a prospective, open-label, multi-centered clinical trial to assess the virologic suppression and immune recovery rates as well as tolerability of the regimen 3TC+TDF+EFV in ARV-naive Chinese population.

500 eligible participants will be recruited to take the regimen If the patient fails to tolerate EFV, it can be substituted by NVP when CD4 < 250/μL, and by LPV/r when CD4 > 250/uL. If the patient fails to tolerate TDF, AZT will be an alternative, except when Hb < 90/L or neutrophil count < 0.75×109/L. The participants will be followed up by months 0.5, 1, 2 ,3 and every 3 months subsequently for 2 years.

The efficacy of the regimen will be evaluated by comparison between different points along the time line and previous regimens. The safety of the regimen will be assessed by monitoring kidney function, bone density, cardiovascular profile, lipid profile, liver function etc as well as other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65 years of either gender
* HIV-1 antibody seropositive detected by ELISA and confirmed by western blot
* CD4 cell count < 500/ul
* Signed informed consent, with no condition that precludes follow-up for 2 years
* No plan to move out of the area during the trial
* antiretroviral therapy naive

Exclusion Criteria:

* patients in acute phase of HIV infection
* patients with ongoing opportunistic infection or AIDS-related malignancies; or with opportunistic infection within previous 3 months and still unstable within 14 days before inclusion
* patients with the any of the following test results during screening for inclusion:

  * WBC count < 2000/ul,
  * neutrophil count < 1000/ul,
  * Hb < 9g/dl,
  * platelet count < 75000/ul,
  * serum creatinine > 1.5 ULN,
  * transaminases or alkaline phosphatase > 3 ULN,
  * total bilirubin > 2 ULN,
  * serum creatinine kinase > 2 ULN
* CCr < 60ml/min
* Pregnancy and breastfeeding
* Intravenous drug user
* Severe neuropathy or mental disorder
* history of alcohol abuse and unable to withdrawal
* Severe peptic ulcer disease
* Non-Chinese nationality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 48 | 48 weeks

SECONDARY OUTCOMES:
Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 96 | 96 weeks
Percentage of Participants With HIV-1 RNA < 40 Copies/mL at Week 96 | 96 weeks
Change From Baseline in CD4 count at Week 48 | Baseline and 48 weeks
Change From Baseline in CD4 count at Week 96 | Baseline and 96 weeks
Incidence of adverse events and laboratory abnormalities from baseline to week 48 | 48 weeks
Incidence of adverse events and laboratory abnormalities from baseline to week 96 | 96 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Fan H, Guo F, Hsieh E, Chen WT, Lv W, Han Y, Xie J, Li Y, Song X, Li T. Incidence of hypertension among persons living with HIV in China: a multicenter cohort study. BMC Public Health. 2020 Jun 1;20(1):834. doi: 10.1186/s12889-020-08586-9. PMID 32487185
- [Derived] Luo L, Wang N, Yue Y, Han Y, Lv W, Liu Z, Qiu Z, Lu H, Tang X, Zhang T, Zhao M, He Y, Shenghua H, Wang M, Li Y, Huang S, Li Y, Liu J, Tuofu Z, Routy JP, Li T. The effects of antiretroviral therapy initiation time on HIV reservoir size in Chinese chronically HIV infected patients: a prospective, multi-site cohort study. BMC Infect Dis. 2019 Mar 14;19(1):257. doi: 10.1186/s12879-019-3847-0. PMID 30871484